CLINICAL TRIAL: NCT00734578
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multi-Center, Dose Optimization Study Evaluating the Efficacy and Safety of SPD503 in Combination With Psychostimulants in Children and Adolescents Aged 6-17 Years With a Diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy and Safety of SPD503 in Combination With Psychostimulants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-313
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPD503-AM (Experimental): SPD503 (Guanfacine Extended Release)
  Interventions: Drug: SPD503-AM
- SPD503-PM (Experimental): SPD503 (Guanfacine Extended Release)
  Interventions: Drug: SPD503-PM
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503-AM — SPD503 (Guanfacine Extended Release)-AM Optimized 1-4mg
  Other Names: Intuniv
  Arms: SPD503-AM
Drug: SPD503-PM — SPD503 (Guanfacine Extended Release)-PM Optimized 1-4mg
  Other Names: Intuniv
  Arms: SPD503-PM
Drug: Placebo — Placebo matched to Guanfacine Hydrochloride Extended Release
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of SPD503 in subjects with ADHD when co-administered with psychostimulants in children and adolescents aged 6-17 years with a diagnosis of ADHD with a sub-optimal, partial response to stimulants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with ADHD currently taking a stable dose of psychostimulant for at least 4 weeks
* Aged 6-17 years with a sub-optimal
* Partial response to stimulants
* Subjects must be < 95th percentile for BMI with weight >= 55lbs and <= 176lbs

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 461 (Actual)
Dates: Start 2008-09-02 (Actual); Primary Completion 2009-12-10 (Actual); Study Completion 2009-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (61):
- United States (61):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Melmed Center, Scottsdale, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - UCSD Department of Psychiatry, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Miami Children's Hospital, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - AMR-Baber Research, Inc., Naperville, Illinois
  - American Medical Research, Inc, Oak Brook, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Pedia Research, Newburgh, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Marc Hertzman, MD, PC, Rockville, Maryland
  - Delmarva Family Resources, Salisbury, Maryland
  - Massachussests General Hospital, Cambridge, Massachusetts
  - Neurobehaviorial Medicine, Bloomfield Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Behavioral Medicine Center, Troy, Michigan
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Midwest Research Group/St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Premier Psychiatric Research Inst. LLC, Lincoln, Nebraska
  - Centers for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center ADHD Program, Durham, North Carolina
  - Triangle Neuropsychiatry, PLLC, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Department of Psychiatry, The Ohio State University, Columbus, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc, Eugene, Oregon
  - Oregon Center for Clinical Investigations, INC (OCCI, Inc.), Portland, Oregon
  - Summit Research Network, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Peds Research Inc., Barnwell, South Carolina
  - FutureSearch Trials, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Claghorn-Lesem Research Clinic, Inc., Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Western Clinical Investigations, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Wharton Research Center, Wharton, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - Psychiatric Alliance of the Blue Ridge Clinical Research, Charlottesville, Virginia
  - NeuroScience, Inc, Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Alliance Research Group, Richmond, Virginia
  - Bayou City Research, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Result] Wilens TE, Bukstein O, Brams M, Cutler AJ, Childress A, Rugino T, Lyne A, Grannis K, Youcha S. A controlled trial of extended-release guanfacine and psychostimulants for attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2012 Jan;51(1):74-85.e2. doi: 10.1016/j.jaac.2011.10.012. Epub 2011 Nov 25. PMID 22176941
- [Derived] Cutler AJ, Brams M, Bukstein O, Mattingly G, McBurnett K, White C, Rubin J. Response/remission with guanfacine extended-release and psychostimulants in children and adolescents with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2014 Oct;53(10):1092-101. doi: 10.1016/j.jaac.2014.08.001. Epub 2014 Aug 15. PMID 25245353
- See also: FDA Recall Information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved Label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD503-AM + Psychostimulant: Guanfacine Hydrochloride Extended Release administered in the AM plus a psychostimulant (subject was on a stable dose on entry and maintained throughout) administered each morning. This group received a matching placebo in the PM. An optimal dose of Guanfacine Hydrochloride Extended Release (1-4 mg/day once-daily) is determined for each subject over 5 weeks. The subject is then maintained on this optimal dose for an additional 3 weeks.
- SPD503-PM + Psychostimulant: Guanfacine Hydrochloride Extended Release administered in the PM plus a psychostimulant (subject was on a stable dose on entry and maintained throughout) administered each morning. This group received a matching placebo in the AM. An optimal dose of Guanfacine Hydrochloride Extended Release (1-4 mg/day once-daily) is determined for each subject over 5 weeks. The subject is then maintained on this optimal dose for an additional 3 weeks.
- Placebo + Psychostimulant: Placebo was administered in both the AM and PM plus a psychostimulant (subject was on a stable dose on entry and maintained throughout) each morning.
Period: Overall Study
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Started | 154 | 153 | 154
Completed | 121 | 128 | 129
Not Completed | 33 | 25 | 25
Not completed — Adverse Event | 4 | 6 | 1
Not completed — Protocol Violation | 8 | 6 | 3
Not completed — Withdrawal by Subject | 7 | 8 | 11
Not completed — Lost to Follow-up | 9 | 3 | 5
Not completed — Lack of Efficacy | 3 | 2 | 5
Not completed — Randomized in error | 1 | 0 | 0
Not completed — Exclusion criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant | Total
Number analyzed (Participants) | 150 | 152 | 153 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] — The demographics are based on the Safety Population (n = 455) which includes all subjects who received at least 1 dose of study drug.
  years | 11.0 (2.6) | 10.6 (2.3) | 10.8 (2.3) | 10.8 (2.4)
Age, Customized [Count of Participants; unit: Participants] — The demographics are based on the Safety Population (n = 455) which includes all subjects who received at least 1 dose of study drug.
  Participants
    6-17 years | 150 | 152 | 153 | 455
Sex: Female, Male [Count of Participants; unit: Participants] — The demographics are based on the Safety Population (n = 455) which includes all subjects who received at least 1 dose of study drug.
  Participants
    Female | 42 | 46 | 41 | 129
    Male | 108 | 106 | 112 | 326
Region of Enrollment [Count of Participants; unit: Participants] — The demographics are based on the Safety Population (n = 455) which includes all subjects who received at least 1 dose of study drug.
  Participants
    United States | 150 | 152 | 153 | 455

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at Week 8 - Last Observation Carried Forward (LOCF)
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and weekly up to 8 weeks
Population: Full Analysis Set (FAS) which includes all subjects who received at least 1 dose of any study drug during this study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 148 | 152
Units on a scale | -20.4 (12.77) | -21.0 (12.39) | -16.0 (11.77)
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; The null hypothesis stated that there was no difference between SPD503 AM or placebo and that there was no difference between SPD503 PM or placebo. 90% power was needed to detect an effect size of at least 0.4 between either SPD503 group and placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — Both SPD503 groups were compared with placebo using Dunnett's adjustment. Each treatment comparison was evaluated at the 0.05 significance level (Dunnett's adjusted); Placebo-adjusted difference in LS mean = -4.5, 95% CI [-7.5 to -1.4]
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Placebo-adjusted difference in LS mean = -5.3, 95% CI [-8.3 to -2.3]

2. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) at Week 8 - LOCF
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 148 | 152
Percent of participants | 70.5 | 74.3 | 57.9
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.024, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons

3. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S) at Week 8 - LOCF
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 148 | 152
Percent of participants
  Normal, not at all ill | 22.8 | 25.0 | 15.1
  Borderline mentally ill | 19.5 | 26.4 | 17.8
  Mildly ill | 34.2 | 26.4 | 28.9
  Moderately ill | 16.1 | 16.2 | 27.0
  Markedly ill | 6.0 | 5.4 | 9.2
  Severely ill | 1.3 | 0.7 | 2.0
  Most extremely ill | 0.0 | 0.0 | 0.0
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.013, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons

4. Secondary Outcome: Change From Baseline in Conners' Global Index - Parent (CGI-P) Total Score at Week 8 - LOCF: Morning Assessment (Before School)
Description: The index contains 10 items. Each item on the scale is scored from a range of 0 (reflecting never, seldom) to 3 (reflecting very often, very frequent) with total scores ranging from 0 to 30.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 147 | 153
Units on a scale | -8.4 (7.27) | -9.6 (7.68) | -6.9 (6.89)
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.019, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -1.7, 95% CI [-3.2 to -0.3]
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -2.6, 95% CI [-4.0 to -1.1]

5. Secondary Outcome: Change From Baseline in Conners' Global Index - Parent (CGI-P) Total Score at Week 8 - LOCF: Evening Assessment (Before Bedtime)
Description: The index contains 10 items. Each item on the scale is scored from a range of 0 (reflecting never, seldom) to 3 (reflecting very often, very frequent) with total scores ranging from 0 30.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 147 | 153
Units on a scale | -8.2 (7.79) | -8.8 (7.21) | -6.0 (6.84)
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.002, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -2.4, 95% CI [-4.0 to -0.9]
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -3.0, 95% CI [-4.5 to -1.5]

6. Secondary Outcome: Percentage of Participants With Improvement on Parent Global Assessment (PGA) at Week 8 - LOCF
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: Baseline and week 8
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 129 | 133 | 141
Percent of participants | 69.8 | 67.7 | 47.5
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons

7. Secondary Outcome: Change From Baseline in the Oppositional Subscale of the Conners' Parent Rating Scale-Revised Long Form (CPRS-R:L) Score at Week 8 - LOCF
Description: The oppositional subscale of the CPRS-R:L contains 10 items designed to reflect criteria for oppositional defiance disorder (ODD). Each item is scored on a range from 0 (not true at all) to 3 (very much true) with total scores ranging from 0 to 30. Higher scores are reflective of more severe symptoms.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 129 | 134 | 141
Units on a scale | -6.6 (6.97) | -6.3 (7.05) | -4.2 (6.79)
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.001, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -2.4, 95% CI [-3.9 to -0.9]
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.003, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -2.2, 95% CI [-3.6 to -0.7]

8. Secondary Outcome: Change From Baseline in Before School Functioning Questionnaire (BSFQ) at Week 8 - LOCF
Description: This scale was designed to assess symptoms of ADHD that typically occur in the morning. The BSFQ consists of two components. The first, a 20-item scale with ratings from 0 (none) to 3 (severe) with a range of 0-60 followed by two questions answered with duration of time (in minutes). The second, a 14-item scale with ratings from 0 (no) to 2 (a lot) with a range of 0-28. The results reported here are from the 20-item scale. Lower scores are better.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 141 | 141 | 144
Units on a scale | -16.7 (13.87) | -16.7 (13.45) | -11.5 (13.45)
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p < 0.001, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -5.1, 95% CI [-8.0 to -2.2]
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.002, ANCOVA — No adjustments for multiple comparisons; Placebo-adjusted difference in LS mean = -4.7, 95% CI [-7.6 to -1.7]

9. Secondary Outcome: Post Sleep Questionnaire (PSQ) Quality of Sleep at Week 8 - LOCF
Description: Post Sleep Questionnaire (PSQ) overall rating of quality of sleep. There are 5 rating responses ranging from very poor to very good. No numbers are associated with the rating responses.
Time Frame: Baseline and weekly up to 8 weeks
Population: FAS
Measure: Number; unit: Percent of participants
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Number analyzed (Participants) | 149 | 148 | 153
Percent of participants
  Very poor | 0.7 | 0.7 | 0.0
  Poor | 6.7 | 6.8 | 3.3
  Average | 26.8 | 29.7 | 33.3
  Good | 40.3 | 41.2 | 40.5
  Very good | 25.5 | 21.6 | 22.9
Statistical Analysis 1: Comparison: SPD503-AM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.971, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: SPD503-PM + Psychostimulant vs Placebo + Psychostimulant; Not powered for secondary outcome measures; Test type: Superiority or Other; p = 0.502, Cochran-Mantel-Haenszel — No adjustments for multiple comparisons

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: For the serious adverse events: syncope occurred in the context of nausea, vomiting and sinusitis; self-injurious behavior, aggression, homicidal ideation, and adjustment disorder with mixed disturbance of emotions and conduct in a subject with similar behaviors prior to study start; exposure to toxic agent was poison ivy.
Arm/Group | SPD503-AM + Psychostimulant | SPD503-PM + Psychostimulant | Placebo + Psychostimulant
Serious Adverse Events (participants affected / at risk) | 1/150 | 2/152 | 0/153
Other Adverse Events (participants affected / at risk) | 116/150 | 116/152 | 97/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503-AM + Psychostimulant (N=150) | SPD503-PM + Psychostimulant (N=152) | Placebo + Psychostimulant (N=153)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Self injurious behavior (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503-AM + Psychostimulant (N=150) | SPD503-PM + Psychostimulant (N=152) | Placebo + Psychostimulant (N=153)
Headache (Nervous system disorders) | 32 | 32 | 20
Somnolence (Nervous system disorders) | 21 | 20 | 7
Upper respiratory tract infection (Infections and infestations) | 14 | 16 | 12
Nausea (Gastrointestinal disorders) | 4 | 11 | 5
Fatigue (General disorders) | 18 | 11 | 4
Insomnia (Psychiatric disorders) | 8 | 18 | 6
Abdominal pain upper (Gastrointestinal disorders) | 12 | 13 | 3
Dizziness (Nervous system disorders) | 15 | 8 | 6
Decreased appetite (Metabolism and nutrition disorders) | 9 | 11 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 7
Irritability (General disorders) | 6 | 9 | 11
Pyrexia (General disorders) | 6 | 8 | 6
Sedation (Nervous system disorders) | 5 | 8 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.